CLINICAL TRIAL: NCT07033208
Title: Feasibility of a Wireless Thermal Capsule Endoscopy to Detect Gastrointestinal Thermal Variance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator - MD, PhD, FACC, FCAP, FNAI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2023P002565
Record Dates: First submitted 2025-05-02; First posted 2025-06-24 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Healthy
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy Volunteers (Experimental): 10 healthy adult participants with no pre-existing gastrointestinal disorders will be enrolled at MGH
  Interventions: Device: Feasibility to obtain thermal variance measurements using a wireless thermal capsule

INTERVENTIONS:
Device: Feasibility to obtain thermal variance measurements using a wireless thermal capsule — A total of 10 healthy participants will be enrolled in this study all consented participants will receive the same intervention.

SUMMARY:
The goal of this research is to learn how a new device called the wireless thermal capsule (WTC) can collect thermal data to help see diseases that happen in the gastrointestinal (GI) tract, such as Crohn's Disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of using the wireless thermal capsule (WTC) to collect temperature information from the human GI tract in healthy adult subjects. Participants will be asked to do a standard of care bowel prep with instructions to start the prep three days before their scheduled procedure. Participants may also be asked to fast for several hours and consume a series of laxative prep mixtures. Participants will be given a bed to sit in the Translational and Clinical Research Center at MGH. After informed consent, a receiver belt and 8 antennas will be placed on the subjects abdomen by trained study staff. The participant will be asked to swallow the WTC capsule, and will have 10 attempts to try to swallow the capsule. They may be also offered optional swallowing aids such as PillGlide or Chloraseptic to help swallow the capsule. If the participant is not able to swallow the capsule after 10 attempts, the research procedure will be terminated. Once the WTC has been swallowed, the research study team will monitor the subject hourly and collect thermal and position tracking data from the WTC as it travels the GI tract and is excreted in their stools. The participant will be asked to stay for up to 16 hrs or until the capsule has been passed, which ever is earlier. Should the participant experience any new symptoms that could indicate a problem in the GI tract, (abdominal discomfort, blood in stool, nausea), a physician will be consulted. The participant may be asked to consume drugs such as metoclopramide or polyethylene glycol to help move the capsule along in their gut. If the capsule hasn't been passed after 16 hours, the participant may be cleared to return home if they have no other symptoms, and may be asked to self monitor until the capsule has passed. The study team will follow up with the participant until the capsule has passed, and the participant may be asked to provide visual confirmation that the capsule has been successfully passed at home. If passage is not confirmed after 2 weeks, the participant may be asked to return to MGH for medical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 -75 years old
* Participant is considered healthy, with no known illnesses
* Participant can follow fasting requirements
* Participant can follow bowel prep instructions
* Participant can provide informed consent

Exclusion Criteria:

* Participant is older than 75 years of age
* Participant with current dysphagia or any swallowing disorder
* Participant with any current condition believed to have an increased risk of capsule retention such as gastrointestinal strictures, intestinal tumors, bowel obstruction, incomplete colonoscopies or fistula
* Participant with a diagnosis of gastroparesis or small bowel or large bowel dysmotility
* Participant with a history of inflammatory bowel disease (IBD), intestinal Crohn's disease, chronic constipation, or rectal bleeding
* Participant with clinical evidence of renal disease, including clinically significant laboratory abnormalities of renal function within the past 6 months
* Participant with chronic usage of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Participants with a known contradiction to metoclopramide
* Participants with a known contraindication to polyethylene glycol
* Participant with currently suspected or diagnosed with hematochezia, melena, iron deficiency with or without anemia
* Participant who has had intestinal surgery in the past
* Participant with a history of congestive heart failure
* Participant with Type I or Type II Diabetes
* Participant has a cardiac pacemaker or other implanted electromedical device.
* Participant expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Participant has participated in an investigational drug or device research study within 30 days of enrollment that may interfere with the subject's safety or ability to participate in this study
* Participant with delayed gastric emptying
* Participant who is pregnant, suspected pregnant, or is actively breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Gastrointestinal Temperature Mean Variance in adult study participants as measured by the wireless thermal capsule | 2 weeks
  This is a pilot study to demonstrate that the capsule can transmit valid temperature data from within the gastrointestinal tract. Since the study participants are nominally healthy, we anticipate that on a per patient basis, the capsule will detect a core body temperature with a mean variance (σ^2) of +/- 0.5°C. With a study size of 10 participants, the measured mean variance 95% confidence intervals will be 0.24≤σ^2≤1.6 °C, which is sufficient to demonstrate that the capsule transmits valid gastrointestinal tract temperature data.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No